CLINICAL TRIAL: NCT03677310
Title: The Effects of 3% Sodium Chloride on Post-operative Dysphagia in Patients Undergoing Anterior Cervical Discectomy and Fusion: a Prospective, Randomized Double-blind Trial
Brief Title: Effects of 3% Sodium Chloride on Post-operative Dysphagia Following Anterior Cervical Spine Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Resident physician decided not to proceed with study
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012482
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: There is no effective treatment for post-operative dysphagia. Thus crossover is not expected.
Who Masked: Participant, Investigator
Masking Description: The bags of IV solution will be masked by the pharmacists before sending to the operating room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3% sodium chloride (Experimental): Subjects in this group will receive 3% sodium chloride over a period of 24 hours at a rate of 10 cc/hour beginning immediately prior to incision.
  Interventions: Drug: 3% Sodium Chloride
- Normal Saline (Sham Comparator): This group will receive normal saline over a period of 24 hours at a rate of 10 cc/hour beginning immediately prior to incision.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: 3% Sodium Chloride — 3% sodium chloride will be given intravenously at a rate of 10 cc/hour over a period of 24 hours beginning immediately prior to incision.
  Arms: 3% sodium chloride
Drug: Normal Saline — Normal Saline will be given intravenously at a rate of 10 cc/hour over a period of 24 hours beginning immediately prior to incision.
  Arms: Normal Saline

SUMMARY:
Post-operative dysphagia is a significant issue following anterior cervical spine surgery. The investigators are studying the effects of perioperative 3% sodium chloride, given over a period of 24 hours, on post-operative dysphagia. The goal is to reduce the incidence and severity of post-operative dysphagia.

DETAILED DESCRIPTION:
Based on a priori analysis the investigators will need 100 subjects in a placebo arm (normal saline) and 100 subjects in a treatment arm (3% sodium chloride), for a total of 200 patients. This study will be conducted on healthy subjects with normal renal function undergoing anterior cervical discectomy and fusion for degenerative indications only. Subjects will be randomized to the treatment or placebo arm (which will be double blinded). Subjects in the treatment arm will begin to receive intravenous 3% sodium chloride before the incision is made. The solution will be given at a rate of 10 cc/hour over a period of 24 hours. Baseline, post-operative, and delayed post-operative dysphagia surveys will be administered either in person or by telephone. The investigators hope to decrease the incidence and severity of post-operative dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing anterior cervical discectomy and fusion for degenerative indications

Exclusion Criteria:

* history of cervical trauma
* baseline dysphagia
* age less than 18 years old
* history of previous anterior neck surgery
* Creatinine clearance less than 30
* Creatinine greater than 1.0
* baseline sodium greater than 145
* patients with known electrolyte abnormalities
* congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative dysphagia | Change in dysphagia scores will be assessed from pre-operative baseline value to: post-operative day one value, 2 week value, 6 week value, and 12 week value.
  Dysphagia as assessed by the Bazaz Dysphagia Score. The Bazaz score grades dysphagia based on a short questionnaire as "none", "mild", "moderate", and "severe".

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Tanaka, MD, Principal Investigator — University of Missouri Hospital

IPD SHARING:
Plan to Share IPD: No